CLINICAL TRIAL: NCT01839734
Title: LAMBCHOP-Lubiprostone Activity Among the MicroBiota of the Colon in HIV in Opposing Permeability: Pilot Study of Lubiprostone as a Modulator of Gut Microbial Translocation in HIV With Incomplete CD4 T-cell Recovery on Antiretroviral Therapy
Brief Title: Lubiprostone as a Modulator of Gut Microbial Translocation in HIV With Incomplete CD4 Recovery on Antiretroviral Therapy
Acronym: LAMBCHOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruth M. Rothstein CORE Center (Other)
Responsible Party: Principal Investigator, Gregory Huhn, Attending Physician, Infectious Disease, Ruth M. Rothstein CORE Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-071
Record Dates: First submitted 2013-04-18; First posted 2013-04-25 (Estimated); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: HIV
Keywords: CD4+
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Experimental): 4 weeks of treatment with lubiprostone 24 mcg by mouth (PO) once-daily (Interventional Group)
  Interventions: Drug: Lubiprostone
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Lubiprostone — Lubiprostone 24 mcg by mouth (PO) once-daily
  Other Names: Brand name: Amitiza
  Arms: Lubiprostone

SUMMARY:
The use of lubiprostone will decrease the levels of immune activation in HIV-infected subjects with incomplete CD4+ T-cell recovery with antiretroviral therapy (ART).

* Lubiprostone will decrease levels of translocated gut microbial products in HIV-infected subjects with incomplete CD4+ T-cell recovery with ART.
* The decrease in levels of translocated gut microbial products will be associated with a decline in the levels of immune activation in HIV-infected subjects with incomplete CD4+ T-cell recovery with ART.

DETAILED DESCRIPTION:
Incomplete immune recovery in HIV-infected individuals is associated with impaired immune response to antigens, opportunistic infections, cardiovascular disease and malignancies, and increased mortality. Several studies have pointed to increased microbial translocation and immune activation as playing a causative role in these patients with limited CD4 recovery with antiretroviral therapy (ART). The gut mucosa of HIV-infected individuals sustains a rapid and profound depletion of gut mucosal CD4+ T-cells as early as a few days after infection. These changes lead to defects in mucosal immune and epithelial barrier function that allows the translocation of gut microbial products, such as plasma LPS (endotoxin) and bacterial 16s DNA. Plasma endotoxin and bacterial 16s DNA are elevated in HIV-infected individuals and their levels are associated with increased levels of immune activation. ART does not readily reverse the deficits in gut mucosal CD4+ T-cells. The epithelial barrier composed of tight junction complexes of the GI tract is a major defense that must be breached in order for microbial antigens and enterotoxins expressed by pathogenic bacteria to traverse from the lumen of the intestine to the lamina propria of the GI tract. Given recent data demonstrating increased complications and mortality in HIV-infected individuals despite suppressed viral replication on ART, investigators have proposed that adjunctive therapies aimed at reducing microbial translocation and/or its inflammatory consequences could improve the long-term prognosis of HIV-infected individuals. An intervention that decreases the level of translocated gut microbial products using modulators that act at the mucosal tight junction barrier is a strategy that has not been studied in HIV.

LAMBCHOP is a randomized, open-label, controlled two-arm study that will test whether 4 weeks of treatment with lubiprostone, an apical lumen ClC-2 chloride channel activator licensed for the treatment of chronic idiopathic constipation and irritable bowel syndrome with constipation, reduces levels of translocated gut microbial products and markers of immune activation in HIV-infected subjects on antiretroviral therapy with incomplete CD4 recovery. Lubiprostone is a potent intestinal epithelial secretagogue that has been shown to stimulate recovery of mucosal barrier function via the restoration of tight junction protein complexes in ex vivo studies of ischemic porcine intestine. This study will take advantage of lubiprostone's known effect in vitro to significantly decrease E. coli and S. typhimurium translocation in a concentration-dependent manner and in in vivo mouse studies to promote enhanced protection against translocated pathogenic bacteria by shifting the intestinal microbiota in order to study the role of translocated gut microbial products in driving immune activation in HIV-infected subjects. Blood samples and stool specimens will be collected at several time points during the study to measure markers of cellular activation, inflammation, gut translocation, and coagulation. Safety assessments will be performed at screening, entry, and several post-entry visits. The primary objectives of the study is to determine whether there is a significant difference in levels of immune activation and gut microbiome after 4 weeks of study drug in those who received lubiprostone.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.
* On tenofovir/emtricitabine/efavirenz single tablet combination therapy for at least 72 weeks prior to study entry.
* No plans to change the antiretroviral regimen at least in the next 3 months after study entry.
* CD4+ cell count < 350 cells/mm3 obtained within 120 days prior to study entry at any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
* All previous CD4+ cell counts should be < 350 cells/mm3 for at least 72 weeks prior to study entry while subjects were on ART.
* Documentation of HIV-1 RNA below the limit of detection (e.g., < 50 copies/mL on Roche Amplicor HIV-1 Monitor assay, < 75 copies/mL on the Versant HIV-1 RNA assay by branched DNA, < 400 copies/mL on a standard Roche Amplicor assay, < 40 copies/mL on the Abbott m2000sp/m2000rt real-time PCR test, < 48 copies/mL on the COBAS AmpliPrep/TAQMAN HIV-1 assay) verified by at least two measurements prior to study entry, one of which must be at least 48 weeks prior to study entry and one measurement that was obtained between 121 days and 48 weeks prior to study entry.
* Screening HIV-1 RNA below the limit of detection obtained within 120 days prior to study entry using a FDA -approved assay (e.g., < 50 copies/mL on Roche Amplicor HIV-1 Monitor assay, < 75 copies/mL on the Versant HIV-1 RNA assay by branched DNA, < 40 copies/mL on the Abbott m2000sp/m2000rt real-time PCR test, < 48 copies/mL on the COBAS AmpliPrep/TAQMAN HIV-1 assay).
* Fasting laboratory values obtained within 45 days prior to entry as follows:

  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Hemoglobin ≥ 10.0 g/dL
  * Platelet count ≥ 50,000/mm3
  * International normalized ratio (INR)
* Female subjects of reproductive potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months; i.e., those who have had menses within the preceding 24 months or have not undergone a sterilization procedure [hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or bilateral salpingectomy]) must have a negative serum or urine β-HCG pregnancy test with a sensitivity of at least 50 mIU/mL performed within 24 hours prior to study entry.

If participating in sexual activity that could lead to pregnancy, the female subject must agree to use one form of contraceptive as listed below while receiving protocol-specified treatment and for 4 weeks after stopping the treatment.

* If the female subject is not of reproductive potential (girls who have not reached menarche, women who have been post-menopausal for at least 24 consecutive months, or women who have undergone surgical sterilization, e.g., hysterectomy, bilateral oophorectomy, or bilateral tubal ligation or salpingectomy), she is eligible without requiring the use of a contraceptive. Self report is acceptable documentation of sterilization, other contraceptive methods, and menopause.
* Men and women age ≥ 18 and ≤ 65 years of age.
* Ability and willingness of subject or legally authorized representative to provide informed consent.

Exclusion Criteria:

* Active diarrhea (3 or more unformed stools per day) within 28 days prior to study entry (except if site investigator or primary care provider attributes diarrhea to antiretroviral or azithromycin use).
* History of or active inflammatory bowel disease.
* History of significant liver disease, defined as having chronic liver disease (including chronic alcoholic liver disease, hepatitis B or C), plus either: a) ascites, b) encephalopathy, or c) a Child-Pugh Score of > 7.
* Receipt of antimicrobial therapy within 30 days prior to study entry.

NOTE: Antimicrobial use for prophylaxis of opportunistic infections, e.g., azithromycin or trimethoprim-sulfamethoxazole, is allowed.

* Active infection requiring the use of antibiotics within 30 days prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of study drug or their formulation.
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to entry.
* Use of any of the following medications for more than 3 consecutive days within the 60 days prior to study entry:

  * Immunosuppressives (e.g., azathioprine, corticosteroids [physiologic replacement doses are allowed], cyclosporine, mycophenolate, NSAIDs (nonsteroidal anti-inflammatory drugs), sirolimus, sulfasalazine, tacrolimus)
  * Immune modulators (e.g., cytokines [e.g., IL-2], granulocyte colony stimulating factor, growth hormone, tumor necrosis factor antagonists, thalidomide)
  * Antineoplastic agents
  * Probiotics (defined as products that contain significant amounts of live microorganisms and are ingested for specific health benefits, e.g., yogurt with live and active cultures, Lactobacillus GG, Saccharomyces boulardii)
  * Anticoagulants (e.g., warfarin and heparin)
* Vaccinations within 1 week prior to the pre-entry or study entry visits.

NOTE: Subjects are encouraged to get the flu vaccine prior to study pre-entry visit.

* Participation on any HIV immunotherapy/therapeutic vaccination trials within 6 months prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Huhn, MD, MPHTM, Principal Investigator — Ruth M. Rothstein CORE Center
Locations (1):
- Ruth M. Rothstein CORE Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant at screening was not randomized because they declined
Groups:
- Arm A: 4 weeks of treatment with lubiprostone 24 mcg by mouth (PO) once-daily (Interventional Group)
  Lubiprostone: Lubiprostone 24 mcg by mouth (PO) once-daily
- Arm B: No intervention
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 16 | 4
Completed | 16 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 16 | 4 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [46 to 54] | 49 [40 to 55] | 49 [45 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 13 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gut Microbial Translocation (iFABP)
Description: Summary difference of participant's median iFABP MT marker change at week 4 from baseline aggregate median values
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Lubiprostone: 24 ug once daily for 4 weeks
- Control: No medication
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
pg/mL
  iFABP Baseline | 145.76 [118.14 to 169.35] | 125.36 [82.43 to 267.76]
  iFABP Week 4 | 151.5 [75.86 to 206.63] | 111.73 [98.44 to 139.84]
  iFABP 4 Week summary difference | -9.34 [-74.32 to 71.74] | 14.47 [-155.83 to 43.93]

2. Primary Outcome: Changes in Gut Microbial Translocation (Zonulin)
Description: Summary difference of participant's median Zonulin MT marker change at week 4 from baseline aggregate median values.
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: ng/ML
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
ng/ML
  Zonulin Baseline | 1 [0.95 to 1.11] | 3.24 [1.46 to 7.14]
  Zonulin Week 4 | 1.06 [0.83 to 1.88] | 0.98 [0.77 to 2.04]
  Zonulin 4 Week Summary Difference | 0.05 [-0.08 to 0.15] | -1.80 [-6.16 to 0.37]

3. Primary Outcome: Changes in Gut Microbial Translocation (sCD14)
Description: Summary difference of participant's median sCD14 MT marker change at week 4 from baseline aggregate median values
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
pg/mL
  sCD14 Baseline | 10807.06 [9198.00 to 12183.11] | 12370.30 [9548.08 to 13117.20]
  sCD14 Week 4 | 11177.92 [10025.86 to 12108.48] | 11345.27 [8565.97 to 13704.10]
  sCD14 4 Week Summary Difference | 247.20 [-1499.26 to 2414.21] | -930.48 [-1448.47 to 1053.26]

4. Primary Outcome: Changes in Gut Microbial Translocation (sCD163)
Description: Summary difference of participant's median sCD163 MT marker change at week 4 from baseline aggregate median values
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
pg/mL
  sCD163 Baseline | 73.09 [54.57 to 92.88] | 51.75 [28.68 to 73.13]
  sCD163 Week 4 | 69.96 [50.61 to 94.16] | 56.74 [29.21 to 90.24]
  sCD163 4 Week Summary Difference | -2.56 [-10.39 to 6.81] | 4.99 [0.54 to 17.12]

5. Secondary Outcome: Changes in Systemic Inflammation (IL-6)
Description: Summary difference of participant's median IL-6 inflammation marker change at week 4 from baseline aggregate median values.
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
pg/mL
  IL-6 Baseline | 1.46 [1.11 to 1.66] | 1.72 [1.44 to 6.51]
  IL-6 Week 4 | 1.67 [1.19 to 2.48] | 2.65 [0.75 to 6.64]
  IL-6 4 Week Summary Difference | -0.12 [-0.49 to 0.38] | -0.68 [-1.48 to 0.93]

6. Secondary Outcome: Changes in Systemic Inflammation (hsCRP)
Description: Summary difference of participant's median hsCRP inflammation marker change at week 4 from baseline aggregate median values
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
pg/mL
  hsCRP Baseline | 25.99 [13.97 to 60.57] | 21.48 [4.73 to 48.47]
  hsCRP Week 4 | 27.72 [14.76 to 47.94] | 22.97 [11.53 to 54.39]
  hsCRP 4 Week Summary Difference | 0.51 [-4.98 to 6.17] | 6.80 [-1.47 to 14.19]

7. Secondary Outcome: Changes in Peripheral CD4+
Description: Summary difference of participant's median CD4+ change at week 4 from baseline aggregate median values
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
cells/mm^3
  CD4+ Baseline | 333 [275 to 384.5] | 329.5 [229.5 to 379.5]
  CD4+ Week 4 | 339 [269.5 to 405.5] | 230 [196 to 336]
  CD4+ 4 Week Summary Difference | 5.5 [-27.05 to 24.5] | -17.5 [-107 to 30]

8. Secondary Outcome: Number of Participants With Adverse Events During Study Period
Description: Safety monitoring, defined as Grade ≥ 2 signs and symptoms, Grade ≥ 2 laboratory abnormalities, and other serious adverse events (SAEs) not otherwise specified.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lubiprostone | Control
Number analyzed (Participants) | 16 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- No Intervention: No medication
Arm/Group | Lubiprostone | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/4
Other Adverse Events (participants affected / at risk) | 8/16 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone (N=16) | No Intervention (N=4)
Other adverse events (Gastrointestinal disorders) | 8 (8) | 0 (0) — Soft stools

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes